CLINICAL TRIAL: NCT05818371
Title: Non-invasive Neuromonitoring Through Point-of-care Determination of ONSD and Assessment of Dynamic Properties of the Optic Nerve Sheath in a Neurointensive Care Setting
Brief Title: Non-invasive ONSD-based Neuromonitoring in a Neurointensive Care Setting
Acronym: ONSDDynamics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ONSDTue
Record Dates: First submitted 2023-03-02; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Trauma, Brain; Subarachnoid Hemorrhage; Intracranial Hypertension
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Intracranial Hypertension

STUDY DESIGN:
Intervention Model Description: Single center, prospective, open diagnostic study, proof-of-concept
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pathologic and non-pathologic intracranial pressure (Other): Sonographic determination of Optic nerve sheath. Parallel recording of ICP
  Interventions: Diagnostic Test: Sonographic determination of the optic nerve sheath diameter

INTERVENTIONS:
Diagnostic Test: Sonographic determination of the optic nerve sheath diameter — Ultrasound-based determination of the optic nerve sheath diameter

SUMMARY:
Intensive care patients with established invasive intracranial neuromonitoring due to neurotrauma are subjected to a repeated non-invasive sonographic recording of the optic-nerve-sheath-diameter (ONSD). The recorded images are analyzed through a machine-learning-algorithm and an experienced ultrasound operator. Results are correlated to the parallel recorded intracranial pressure (ICP). The study aims to establish ONSD as a supplementary for raised ICP.

DETAILED DESCRIPTION:
During the intensive care stay, patients with implemented invasive intracranial pressure monitoring will have sonographic recording of the optic nerve sheath (video clip) with a parallel recording of the underlying ICP. The obtained image material is then i) analyzed by a machine-learning algorithm and ii) manually by 2 blinded differently experienced examiners (expert, novice) with respect to the ONSD. For the manual procedure, three individual measurements are made for each eye and the mean value is determined.

Subsequently, the measured values of the two examiners and the automated procedure are correlated with the ICP recorded during the sonographic examination.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic or non-traumatic (e.g. SAH) brain injury
* Established invasive intracranial pressure monitoring (either intraparenchymal or Intraventricular)

Exclusion Criteria:

* Soft tissue damage to orbital or periorbital region
* Fracture of the Orbita
* Status post decompressive craniectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Sonographic monitoring of optic nerve sheath | Single measurement post-trauma up to day 10
  Repeated ultrasound-based measurement of optic nerve sheath in millimeter (mm)

SECONDARY OUTCOMES:
Invasively measured intracranial pressure | Continuously from time of admission up to day 10
  Continuously recorded invasively (intra-parenchymal, intra-ventricular) determined intracranial pressure (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Tellermann, MD, Principal Investigator — University Hospital of Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No